CLINICAL TRIAL: NCT06063304
Title: Quantitative MRI For Detection And Tracking of Disease Progression Over 2 Years In Early Knee Osteoarthritis Patients & Healthy Volunteers
Brief Title: Quantitative MRI For Detection and Tracking of Knee Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 22IC8098
Record Dates: First submitted 2023-09-08; First posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis
Keywords: Knee Osteoarthritis; Healthy Volunteer; MRI
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: This group consists of healthy volunteers with no history of knee joint pain (refer to inclusion/exclusion criteria for more details). They will be scanned once and their scans will be used as the baseline to compare the early knee osteoarthritis patient data with. 10 healthy volunteers will be recruited.
- Knee Osteoarthritis Patients: This group consists of early knee osteoarthritis patients (refer to inclusion/exclusion criteria for more details). They will be scanned 4 times over a period of 2 years (at enrolment, 6 months, 12 months and 24 months after enrolment) to see how the disease progresses. Their scans will be compared with the baseline healthy volunteer scans to check for any differences in anatomy and tissue properties. 60 knee osteoarthritis patients will be recruited.

SUMMARY:
The goal of this observational study is to develop whole-joint quantitative MRI techniques that aid in the detection and tracking of osteoarthritis disease progression at 3T and 7T MRI scanners. The research objectives are:

1. Compare the relative accuracies of 7T and 3T MRI in detecting clinical osteoarthritis progression.
2. Compare the quantitative MRI measures developed with the results acquired from the following two questionnaires: Knee Injury and Osteoarthritis Outcome Score (KOOS) and the Visual Analogue Score (VAS).
3. Measure the repeatability of 7T and 3T quantitative MRI methods developed in whole-joint knee imaging
4. Optimize the quality and efficiency of 7T and 3T whole-joint knee MRI

Participants will be scanned at the 3T scanner at the Clinical Imaging Facility at Hammersmith Hospital and/or the 7T scanner at the LOCUS Center at St Thomas' Hospital. Knee osteoarthritis volunteers will be asked to fill out two questionnaires and will be scanned 4 times over a 2 year period (at enrolment, after 6 months, after 12 months and after 24 months) while healthy volunteers will be scanned once at enrolment. Both healthy volunteers and knee osteoarthritis patients will be asked to fill out MRI safety forms before entering the scanner room, and both groups will be scanned up to 90 minutes during each session.

Researchers will compare knee osteoarthritis patients with healthy volunteers to see how their knee anatomy and tissue properties differ.

ELIGIBILITY:
Inclusion Criteria For Healthy Volunteers:

* All people between 40 to 70 years of age
* All people with no history of knee injury, surgery, or knee pain

Exclusion Criteria For Healthy Volunteers:

* Patients with body mass index of more than 35, or body geometry that prevents scanning due to MRI scanner bore width or knee coil diameter
* Patients with varus or valgus malalignment
* Patients with contraindications to MRI
* Patients lacking capacity to consent
* Patients who are pregnant or breast-feeding
* Patients who are participating in a clinical trial(s) for new drugs and/or therapies

Inclusion Criteria for Knee Osteoarthritis Patients:

* All patients with primary osteoarthritis (grade 2-3 per Kellgren-Lawrence Scale)
* Patients who have had radiographs taken as part of their routine clinical care agreed with their orthopaedic surgeon, Mr Gareth Jones. Note that their radiographs must have been acquired a maximum of three weeks from the first, baseline scanning session. This radiograph will be used to check if patients have primary osteoarthritis.
* All patients between 40 to 70 years of age

Exclusion Criteria for Knee Osteoarthritis Patients

* Patients with body mass index of more than 35, or body geometry that prevents scanning due to MRI scanner bore width or knee coil diameter
* Patients with varus or valgus malalignment of more than 5°
* Patients with radiographic osteoarthritis (grade ≥4 per Kellgren-Lawrence Scale, obtained from radiographs)
* Patients with contraindications to MRI
* Patients lacking capacity to consent
* Patients who are pregnant or breast-feeding
* Patients who are participating in a clinical trial(s) for new drugs and/or therapies

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The research team will be recruiting both healthy volunteers and early knee osteoarthritis patients using the inclusion and exclusion criteria detailed above.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of cartilage thickness values at 3T and 7T as a measure of knee osteoarthritis at enrolment, after 6 months, after 12 months and after 24 months | at enrolment, after 6 months, after 12 months and after 24 months
  The cartilage thickness values will be calculated from the MRI scans that will be acquired.

SECONDARY OUTCOMES:
Reproducibility of microstructure maps at 3T and 7T as a measure of knee osteoarthritis at enrolment, after 6 months, after 12 months and after 24 months | at enrolment, after 6 months, after 12 months and after 24 months
  The microstructure maps will be calculated from the MRI scans that will be acquired.
Reproducibility of MOAKS analysis at 3T and 7T as a measure of knee osteoarthritis at enrolment, after 6 months, after 12 months and after 24 months | at enrolment, after 6 months, after 12 months and after 24 months
  MRI Osteoarthritis Knee Score (MOAKS) values will be calculated from the MRI scans that will be acquired. MOAKS is a semi-quantitative scoring tool that scores sub-regions of articular cartilage and bone marrow lesions. Different grades are used to score each sub-region. For cartilage sub-region loss, grade 0 indicates no loss and grade 3 indicates over 75% loss.
Calculate and compare the longitudinal changes in cartilage thickness at 3T and 7T over the 2 year period | at enrolment, after 6 months, after 12 months and after 24 months
  Cartilage thickness will be calculated for scans acquired at the various time points on the 3T and 7T scanners and compared with each other to investigate the change in thickness over the specified time frame.
Calculate and compare the longitudinal changes in microstructure maps at 3T and 7T over the 2 year period | at enrolment, after 6 months, after 12 months and after 24 months
  Microstructure maps will be calculated for scans acquired at the various time points on the 3T and 7T scanners and compared with each other to investigate the change in thickness over the specified time frame.
Calculate minimum detectable effect size for osteoarthritis progression at 3T and 7T with cartilage thickness | at enrolment, after 6 months, after 12 months and after 24 months
Calculate minimum detectable effect size for osteoarthritis progression at 3T and 7T with microstructure maps | at enrolment, after 6 months, after 12 months and after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Neal K Bangerter, PhD, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD with other researchers.